CLINICAL TRIAL: NCT01056172
Title: A Prospective Randomized, Open Labeled, Phase IV, Multicenter Study for Peginterferon Alfa-2a and Weight-based Ribavirin for 16 or 24 Weeks in genotype2 Chronic Hepatitis C Patients Who Achieved Rapid Virologic Response
Brief Title: PegIFN Alfa-2a and RBV for 16 or 24 Weeks in Patients With Chronic Hepatitis C(CHC) 2 With Rapid Virologic Response(RVR)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Severance Hospital (Other); Pusan National University Hospital (Other); Incheon St.Mary's Hospital (Other); Soon Chun Hyang University (Other); Inje University (Other); Inje University Ilsan Paik Hospital (Other); Inje University Haeundae Paik Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Yoon, Assistant Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNUYH-CHC001
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Genotype 2; Rapid virologic response; Sustained virologic response; Peginterferon alfa-2a; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. 24 weeks in RVR patients. (Active Comparator): Peginterferon alfa-2a and weight-based ribavirin (800-1200mg/day) for 24 weeks in patients with RVR.
  Interventions: Drug: Peginterferon alfa-2a and Ribavirin
- B. 16 weeks in RVR patients. (Experimental): Peginterferon alfa-2a and weight-based ribavirin (800-1200mg/day) for 16 weeks in patients with RVR.
  Interventions: Drug: Peginterferon alfa-2a and Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a and Ribavirin — 1. PegIFN alfa-2a (PEgasys) 180 ug/week
  2. Weight-based ribavirin (<65kg: 800mg/day, 65-85kg: 1000mg/day, >85kg: 1200mg/day)
  3. Treatment duration: 16 weeks
  Arms: B. 16 weeks in RVR patients.
Drug: Peginterferon alfa-2a and Ribavirin — 1. PegIFN alfa-2a (PEgasys) 180 ug/week
  2. Weight-based ribavirin (<65kg: 800mg/day, 65-85kg: 1000mg/day, >85kg: 1200mg/day)
  3. Treatment duration: 24 weeks
  Arms: A. 24 weeks in RVR patients.

SUMMARY:
This study aim to evaluate the non-inferiority of sustained virologic response in peginterferon alfa-2a and weight-based ribavirin for 16 weeks compare with standard treatment duration of 24 weeks in patients who achieved rapid virologic response with genotype 2 CHC.

DETAILED DESCRIPTION:
In recent study (the ACCELERATE trial), treatment with peginterferon alfa-2a and ribavirin (800mg/day) for 16 weeks in patients infected with HCV genotype 2 or 3 result in a lower overall sustained virologic response rate than treatment with the standard 24 weeks regimen. Ribavirin was used as a flat dose (800mg/day) in ACCELERATE trial. But, previous studies which used the weight-based dose of ribavirin (800-1400mg/day) had shown that a treatment duration of 16 weeks was as effective as 24 weeks regimen in HCV genotype 2 patients with a RVR. But, there was too small number of patient enrolled study to argue logically about ACCELERATE trial. In this study, we aimed to confirm the non-inferiority peginterferon alfa-2a and weight-based ribavirin for 16 weeks compare with standard treatment duration of 24 weeks in patients who achieved rapid virologic response with genotype 2 CHC.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years old
2. Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
3. Detectable serum quantitative HCV-RNA
4. HCV genotype 2 (VERSANT HCV Genotype Assay (LIPA))
5. Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin

Exclusion Criteria:

1. Co-infection with hepatitis B and/or human immunodeficiency virus (HIV)
2. History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
3. Decompensated liver disease (Child-Pugh class B or C)
4. Neoplastic disease within 5 years
5. Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
6. Women with ongoing pregnancy or breast feeding
7. Hgb < 11 g/dL in women or < 12 g/dL in men at screening
8. Neutrophil count < 1500 cells/mm3 or platelet count < 90,000 cells/mm3 at screening
9. Serum creatinine level > 1.5 times the upper limit of normal at screening
10. Serum alpha-fetoprotein > 100 ng/mL
11. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
12. History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
13. History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
14. History of a severe seizure disorder or current anticonvulsant use
15. Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
16. Inability or unwillingness to provide informed consent or abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 24 weeks post-treatment (week 40 or week 48)

SECONDARY OUTCOMES:
AEs | up to 24 weeks after last treatment visit
  1. 16 weeks treatment arm: 40 weeks
  2. 24 weeks treatment arm: 48 weeks
laboratory parameters | up to 24 weeks after last treatment visit
  1. 16 weeks treatment arm: 40 weeks
  2. 24 weeks treatment arm: 48 weeks
vital signs | up to 24 weeks after last treatment visit
  1. 16 weeks treatment arm: 40 weeks
  2. 24 weeks treatment arm: 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Yoon, M.D, Principal Investigator — Pusan National University Yangsan Hospital
Locations (8):
- South Korea (8):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Pusan National University Hospital, Busan
  - Inje University Pusan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Inje University Ilsan Paik Hospital, Goyang
  - Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Seoul